CLINICAL TRIAL: NCT05123573
Title: Self-Perceived Competence in Mexican Medical Students Undergoing Distance Learning During the COVID-19 Pandemic
Brief Title: Self-Perceived in Medical Students Undergoing Distance Learning
Acronym: SPMSUDL
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator D, Instituto Mexicano del Seguro Social
Other Study IDs: Self-Perceived Competence
Record Dates: First submitted 2021-10-21; First posted 2021-11-17 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Educational Problems; Medical Students; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Clinical Competence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Clinical Skills — evaluate the students' ability to demonstrate essential clinical skills, clinical reasoning and problem-solving skills, management of life-threatening medical conditions, management of common medical problems, and placing the patients' needs and safety at the center of the care process.

SUMMARY:
Our primary objective is identifying the degree of self-perceived competence in medical students without clinical rotations during the COVID-19 pandemic to know how prepared the students could be when they are professionals because they lack clinical skills in front of an actual patient and can be affected to be accepted in hospitals because they will have to acquire a phase of training later. Without a clinical rotation, one can be deprived of the essential educational value.The study design is an observational cross-section study in which an anonymous survey will be shared online on Google Forms platform. Students will be asked for their participation; after obtaining verbal and consent, the survey will be distributed using social media groups such as foundation school groups. For this study, the Spanish version of the Self-Perceived Competence scale will be used (REF). This scale is comprised of 21 questions divided into five factors that assess: 1) demonstration of the essential clinical skills, 2) demonstration of clinical reasoning, decision making, and problem-solving skills, 3) management of life-threatening medical conditions, 4) management of common medical problems and 5) placing patients' needs and safety at the center of the care process. Each item has a Likert scale answers of 4 options ranging from "incompetent (1)", "somewhat incompetent (2)", "somewhat.

ELIGIBILITY:
Inclusion Criteria:

* Medical students currently attending college in a distance learning modality.
* > 18 years

Exclusion Criteria:

* Medical professionals and specialists
* university students
* < 18 years
* Medical students currently attending clinical rotations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population will be medical students currently attending college in a distance learning modality.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Essential clinical skills | Day 1
  use the Self-Perceived Competence Scale to evaluate the students' ability to demonstrate essential clinical skills such as obtaining an accurate medical history, performing a complete systematic physical examination, and analyzing clinical data. This section has 4 items with Likert scale answers ranging from "(1) incompetent" to "(4) competent".
Clinical reasoning and problem-solving skills | Day 1
  use the Self-Perceived Competence Scale to evaluate the students' ability to demonstrate reasoning skills to formulate and prioritize a differential diagnosis, development of management strategies. This section has 2 items with Likert scale answers ranging from "(1) incompetent" to "(4) competent".
Management of life-threatening medical conditions | Day 1
  use the Self-Perceived Competence Scale to evaluate the students' ability to recognize and assess life or organ-threatening conditions. This section has 2 items with Likert scale answers ranging from "(1) incompetent" to "(4) competent".
Management of common medical problems | Day 1
  use the Self-Perceived Competence Scale to evaluate the students' ability to select and apply the most appropriate and cost-effective diagnostic procedures, manage patients with acute and chronic physical and mental problems. This section has 8 items with Likert scale answers ranging from "(1) incompetent" to "(4) competent".
Placing the patients' needs and safety at the center of the care process | Day 1
  use the Self-Perceived Competence Scale to evaluate the students' ability to demonstrate knowledge and skills in the area related to patient safety, analyze the aftermath of medical error, identify and manage clinical risks. This section has 6 items with Likert scale answers ranging from "(1) incompetent" to "(4) competent".

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico